CLINICAL TRIAL: NCT01158976
Title: Impact of Omega-3 Intake During Pregnancy on Maternal Stress and Infant Outcome
Brief Title: Effect of Omega-3 Supplementation During Pregnancy on Regulation of Stress
Acronym: NAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 09-190A; R21HD058269 (NIH)
Record Dates: First submitted 2010-06-28; First posted 2010-07-08 (Estimated); Results first posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Healthy Pregnant Women

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA supplementation (Experimental)
  Interventions: Dietary Supplement: Docosahexanoic Acid
- Soybean Oil (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Docosahexanoic Acid — 450 mg DHA daily beginning at 16-21 weeks gestation and continuing up to time of delivery
  Other Names: Nordic Naturals ProDHA
  Arms: DHA supplementation
Other: Placebo — soybean oils with strawberry flavoring
  Arms: Soybean Oil

SUMMARY:
This will be the first study of the effect of essential fatty acid supplementation in pregnant women living in inner-city poverty on the stress response system during pregnancy. The investigators proposed that essential fatty acid supplementation will be associated with reductions in the experience of stress, more modulated hormonal response to stress, and more optimal regulation of emotion and attention in the infant, even within the context inner-city poverty.

DETAILED DESCRIPTION:
Significance: Pregnant women living in poverty often experience chronic stress, and consequently higher levels of stress hormones. In utero exposure to high levels of stress hormones can negatively affect the developing fetus and later, the infant's capacity for emotion and behavioral regulation. In this proposal we describe a developing program of research designed to reduce the negative impact of prenatal stress on infant health and development via nutritional supplementation of docosahexaenoic acid (DHA) during pregnancy. DHA is a long-chain polyunsaturated fatty acid member of the omega-3 fatty acid family. DHA is found in its highest concentrations in neural cell membranes, affecting receptor function, neurotransmitter uptake, and signal transmission. There is growing evidence that low levels of dietary DHA intake are associated with suboptimal response to stress and that DHA supplementation can modulate stress response. Aims: The goals of the proposed study are to explore whether DHA supplementation during pregnancy is associated with 1) a reduction in maternal perceived stress during pregnancy; 2) a more modulated maternal cortisol response to a stress stimulus during pregnancy, and 3) more optimal regulation of emotion and behavior in the infant. Approach: Sixty-five pregnant women living in inner-city poverty, who consume less than two servings of fish per week, will be randomly assigned to receive 450 mg/daily of DHA or placebo beginning at 16-20 weeks gestation through the end of pregnancy. Perceived stress, pregnancy related stress, stressful life events, anxiety, and depression will be assessed at baseline and at 24, 30, and 36 weeks of pregnancy and at 4 months post-partum. DHA levels will be assessed at baseline and at 36 weeks of pregnancy. Cortisol response to the Trier Social Stress Test will be measured at baseline, 24, and 30 weeks. At 4 months post-partum infant temperament, cognitive development and stress reactivity will be assessed in the laboratory. Investigators: This proposal stems from an National Institute of Mental Health R21 Translational Science Network on prenatal stress and mental health outcomes in the offspring. Three members of that network, Drs. Keenan, Carter, and Glover, are all funded investigators in the area of prenatal stress and child mental health, which is a prioritized area of exploratory research that could directly impact clinical care. They are collaborating on the present application. Innovation: This will be the first randomized controlled study of the effect of DHA supplementation on stress response in pregnant women living in inner-city poverty, and the first study of maternal DHA supplementation on emotion and stress regulation in their infants. Relevance: If DHA supplementation is associated with reductions in perceived stress, more modulated maternal cortisol response to stress, and more optimal emotional and behavioral regulation in the infant, even within the context inner-city poverty, then a comprehensive program of research on the mechanisms by which these associations evolve and the potential for broad-based prevention of poor developmental outcomes among children born to women living in poverty can be launched.

ELIGIBILITY:
Inclusion Criteria:

* African American race
* age between 20 and 34 years
* 16-21 weeks gestation
* household receipt of public assistance (e.g., Medicaid insurance) due to -low-income
* low levels of DHA consumption as defined as less than two fish servings per week.

Exclusion Criteria:

* known medical complications (e.g., gestational diabetes, pre-eclampsia), -regular use of steroid medications
* alcohol use
* cigarettes or use of illegal substances (by maternal report)
* use of blood thinners or anti-coagulants
* use of psychotropic medications
* Body Mass Index >40
* allergy to iodine and/or soy.

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Keenan K, Hipwell AE, Bortner J, Hoffmann A, McAloon R. Association between fatty acid supplementation and prenatal stress in African Americans: a randomized controlled trial. Obstet Gynecol. 2014 Dec;124(6):1080-1087. doi: 10.1097/AOG.0000000000000559. PMID 25415158

RESULTS

PARTICIPANT FLOW:
Groups:
- DHA Supplementation: Docosahexanoic Acid (DHA): 450 mg DHA daily beginning at 16-21 weeks gestation and continuing up to time of delivery
Period: Overall Study
Arm/Group | DHA Supplementation | Soybean Oil
Started | 43 | 21
Completed | 34 | 17
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DHA Supplementation | Soybean Oil | Total
Number analyzed (Participants) | 43 | 21 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 21 | 64
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 21 | 64
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 43 | 21 | 64
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 21 | 64

OUTCOME MEASURES:

1. Primary Outcome: Maternal Cortisol Levels
Description: Maternal stress regulation at 30 weeks gestation
Time Frame: Baseline (pre-stressor)
Population: The analysis population reflects those participants who received treatment and with available data for the cortisol assessment
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 33 | 17
ug/dL | 0.28 (0.20) | 0.34 (0.12)

2. Primary Outcome: Maternal Cortisol Levels
Description: Maternal stress regulation at 30 weeks gestation
Time Frame: 20 minutes post-stressor
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 33 | 17
ug/dL | 0.29 (0.12) | 0.24 (0.12)

3. Primary Outcome: Maternal Cortisol Levels
Description: Maternal stress regulation at 30 weeks gestation
Time Frame: 45 minutes post stressor
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 33 | 17
ug/dL | 0.22 (0.10) | 0.23 (0.14)

4. Primary Outcome: Infant Cortisol Levels
Description: Infant cortisol response to the Still-Face paradigm before stressor
Time Frame: 4 months post-partum
Population: The analysis population reflects those infants whose mothers who received treatment and with available data for the cortisol assessment
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 34 | 15
ug/dL | 0.23 (0.23) | 0.29 (0.28)

5. Primary Outcome: Infant Cortisol Levels
Description: Infant cortisol response to the Still-Face paradigm 20 minutes post-stressor
Time Frame: 4 months post-partum
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 38 | 17
ug/dL | 0.22 (0.15) | 0.32 (0.27)

6. Primary Outcome: Infant Cortisol Levels
Description: Infant cortisol response to the Still-Face paradigm 45 mins post-stressor
Time Frame: 4 months post-partum
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 38 | 17
ug/dL | 0.21 (0.17) | 0.31 (0.20)

7. Secondary Outcome: Maternal Depression Symptoms
Description: Maternal depression symptoms at 16 to 24 weeks gestation, as measured by the Edinburgh Postnatal Depression Scale, a 10-item measure designed to assess pre- and postnatal depression.
  Maximum score: 30 Minimum score: 0 Possible Depression: 10 or greater Mothers who score above 13 are likely to be suffering from a depressive illness of varying severity.
Time Frame: 16-21 weeks gestation
Population: The analysis population reflects those participants who received treatment and with available data for the assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 43 | 20
units on a scale | 13.05 (5.3) | 12.80 (4.2)

8. Secondary Outcome: Maternal Depression Symptoms
Description: Maternal depression symptoms at 24 weeks gestation as measured by the Edinburgh Postnatal Depression Scale, a 10-item measure designed to assess pre- and postnatal depression.
  Maximum score: 30 Minimum score: 0 Possible Depression: 10 or greater Mothers who score above 13 are likely to be suffering from a depressive illness of varying severity.
Time Frame: 24 weeks
Population: The analysis population reflects those participants who received treatment and with available data for the assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 35 | 18
units on a scale | 13.3 (5.1) | 12.11 (4.1)

9. Secondary Outcome: Maternal Depression Symptoms
Description: Maternal depression symptoms at 30 weeks gestation, as measured by the Edinburgh Postnatal Depression Scale, a 10-item measure designed to assess pre- and postnatal depression.
  Maximum score: 30 Minimum score: 0 Possible Depression: 10 or greater Mothers who score above 13 are likely to be suffering from a depressive illness of varying severity.
Time Frame: 30 weeks gestation
Population: The analysis population reflects those participants who received treatment and with available data for the assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 34 | 17
units on a scale | 12.12 (4.8) | 11.35 (5.1)

10. Secondary Outcome: Maternal Perceived Stress Scale (PSS) Score
Description: Perceived stress as measured by the Perceived Stress Scale (Cohen et al, 1983) at baseline. There are 10 questions in this scale and they all refer to typical life stressors.
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress
Time Frame: Baseline: 16 - 21 weeks
Population: The analysis population reflects those participants who received treatment and with available data for the assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 43 | 20
units on a scale | 27.77 (2.2) | 29 (2.7)

11. Secondary Outcome: Maternal Perceived Stress Scale Score
Description: Perceived stress as measured by the Perceived Stress Scale (Cohen et al, 1983) at 24 weeks gestation.
  There are 10 questions in this scale and they all refer to typical life stressors.
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress
Time Frame: 24 weeks gestation
Population: The analysis population reflects those participants who received treatment and with available data for the assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 35 | 18
units on a scale | 28.06 (3.5) | 27.72 (2.0)

12. Secondary Outcome: Maternal Perceived Stress Scale Score
Description: Perceived stress as measured by the Perceived Stress Scale (Cohen et al, 1983) at 30 weeks gestation.
  There are 10 questions in this scale and they all refer to typical life stressors.
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress
Time Frame: 30 weeks gestation
Population: The analysis population reflects those participants who received treatment and with available data for the assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 34 | 17
units on a scale | 27.47 (3.4) | 29.29 (3.1)

13. Secondary Outcome: Infant Birth Weight
Description: Weight of infant
Time Frame: Time of birth, total sample range: 27.60 to 41.60 weeks gestation
Population: The analysis population reflects those infants of participants who received treatment and with available data for the assessment
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 34 | 15
grams | 3074.39 (582.34) | 2919.56 (537.74)

14. Secondary Outcome: Percentage of Infants Who Had a 1-minute Apgar Scores of 9
Description: Percentage of infants who had a 1-minute Apgar scores of 9 Sub scores from 5 categories( Breathing effort, Heart rate, Muscle tone, Reflexes, Skin color) are added together Score range: 1-10 A higher score is better where 7,8,9 are normal
Time Frame: Time of birth, total sample range: 27.60 to 41.60 weeks gestation
Population: as for outcome 13
Measure: Number; unit: percentage of infants
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 34 | 15
percentage of infants | 75.8 | 59.1

15. Secondary Outcome: Gestational Age (GA)
Description: Gestational Age at time of birth Total sample range: 27.60 to 41.60 weeks Below 37 considered premature Mothers typically induced after 41 weeks due to increased pregnancy risks after this time
Time Frame: Time of birth, total sample range: 27.60 to 41.60 weeks gestation
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 34 | 15
Weeks | 38.85 (2) | 38.84 (2.06)

16. Secondary Outcome: Infant's Receptive Communication Scaled Score
Description: Scaled Score on Receptive Communication subscale of Bayley Scale for Infant Development that determines how well a child recognizes sounds and how much a child understands spoken words and directions compared to a group of children within the same age range from across the United States. Subscale consists of 49 items. Child'e scaled score is calculated from total raw scores.
  Scaled score range: 1 - 12 Lower scores indicate more developmental delay.
Time Frame: 3 months old
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 34 | 15
units on a scale | 4.88 (2.66) | 4.33 (1.91)

17. Secondary Outcome: Infant's Expressive Communication Scaled Score
Description: Scaled Score for Expressive Communication subscale of Bayley Scale for Infant Development that determines how well a child recognizes sounds and how much a child communicates using sounds, gestures, or words compared to a group of children within the same age range from across the United States. Subscale consists of 48 items. Child'e scaled score is calculated from total raw scores.
  Scaled score range: 2 - 9 Lower scores indicate more developmental delay.
Time Frame: At approximately 3 months of age
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 34 | 15
units on a scale | 6.21 (1.41) | 6.00 (1.89)

18. Secondary Outcome: Infant's Fine Motor Skills Scaled Score
Description: Fine motor skills subscale score from Bayley Scale for Infant Development. Determines how well a child recognizes sounds and how much a child can use his or her hands and fingers to do things compared to a group of children within the same age range from across the United States. Subscale consists of 66 items. Child's scaled score is calculated from total raw scores.
  Scaled score range: 1 - 8 Lower scores indicate more developmental delay.
Time Frame: Approximately 3 months of age
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 34 | 15
units on a scale | 2.38 (1.88) | 2.33 (2.13)

19. Secondary Outcome: Infant's Gross Motor Skills Scaled Score
Description: Infants Gross Motor skills subscale score from Bayley Scale for Infant Development. Determines how well a child well your child can move his or her body compared to a group of children within the same age range from across the United States. Subscale consists of 72 items. Child's scaled score is calculated from total raw scores.
  Scaled score range: 1 - 6 'Lower scores indicate more developmental delay.
Time Frame: Approximately 3 months of age
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DHA Supplementation | Soybean Oil
Number analyzed (Participants) | 34 | 15
units on a scale | 1.65 (1.20) | 1.60 (1.12)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | DHA Supplementation | Soybean Oil
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/21
Other Adverse Events (participants affected / at risk) | 0/43 | 0/21

LIMITATIONS AND CAVEATS:
Small sample size and attrition of participants over time likely affect the reliability of the findings. There may have been some differential selection bias across the two groups. We relied on maternal report of uptake.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No